CLINICAL TRIAL: NCT07341191
Title: A Phase II Study of Sonrotoclax Plus Zanubrutinib in Patients With Relapsed/Refractory Mantle Cell Lymphoma Planned for Standard of Care CAR-T Cell Therapy
Brief Title: Sonrotoclax Plus Zanubrutinib in Patients With Relapsed/Refractory Mantle Cell Lymphoma Planned for Standard of Care CAR-T Cell Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I245
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma
Keywords: CAR-T; Relapsed; Refractory; BTK inhibitor; BCL2 inhibitor
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — zanubrutinib; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib + Sonrotoclax (Experimental)
  Interventions: Drug: Zanubrutinib; Drug: Sonrotoclax; Biological: CAR-T Cell Therapy

INTERVENTIONS:
Drug: Zanubrutinib — assigned at enrollment
Drug: Sonrotoclax — assigned at enrollment
Biological: CAR-T Cell Therapy — Standard of Care

SUMMARY:
The purpose of this study is to evaluate the effects of adding two oral medications (sonrotoclax plus zanubrutinib) to standard of care chimeric antigen receptor (CAR-T) cell therapy in participants with mantle cell lymphoma.

DETAILED DESCRIPTION:
Combining sonrotoclax (a next-generation BCL-2 inhibitor) with zanubrutinib (a selective BTK inhibitor) in mantle cell lymphoma (MCL)-is expected to be driven by strong biologic synergy, complementary mechanisms, and more durable responses without chemotherapy. Patients participating in this study must already be planning, and be eligible for CAR-T cell therapy outside of this protocol. CAR-T will be administered according to local or provincial guidelines.

If a patient decides to take part in this study, the patient will first get zanubrutinib (if not on it before starting the study), then during the induction phase they will get a combination of sonrotoclax (with a ramp-up dosing schedule) plus zanubrutinib followed by CAR-T cell therapy, followed zanubrutinib alone/ maintenance.

After finishing study treatment, and even if patients stop treatment early, the study doctor will continue to follow the patient's condition for the rest of their life or until all study results are known

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed mantle cell lymphoma that is relapsed or refractory after at least one prior line of systemic therapy
* Eligible for and planned to receive Health Canada approved CAR-T.
* Have a formalin fixed paraffin embedded tumour tissue block available and must have provided informed consent for the release of the block.
* Presence of radiologically documented disease.
* Measurable disease (one site bidimensionally measurable).
* Age ≥ 18 years.
* Have an ECOG performance status of 0, 1 or 2
* Anticipated life expectancy of ≥ 6 months
* Adequate hematologic and biochemical parameters
* Must have received prior systemic therapy as shown below;
* At least one line of systemic therapy including a Bruton's Tyrosine Kinase inhibitor (BTKi).
* Participants who have previously received venetoclax, sonrotoclax, or any other BCL2 inhibitor (BCL2i) are eligible as long as progressive disease did not occur within 6 months of the last dose of BCL2i. Participants with progressive disease during BCL2i therapy or within 6 months of last dose are not eligible.
* Participants must enter the study while on a BTKi or enroll to a substudy of the protocol to receive zanubrutinib for a minimum duration prior to enrolling to the main study.
* Participants previously exposed to zanubrutinib are eligible irrespective of response to treatment.
* Participants entering the study while on a BTKi must have their BTKi switched to zanubrutinib supplied through the study.
* Participants must have recovered to ≤ grade 1 from all reversible toxicity related to prior therapies.
* Adequate washout must be followed per protocol.
* Prior high-dose myelosuppresive radiation is permitted ≥28 prior to enrollment.
* Previous major surgery is permitted ≥28 days prior to enrollment. Participants of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria

* • Participants on active anticancer therapy for other advanced or metastatic malignancies.
* Concurrent treatment with other anti-cancer therapy
* Serious illnesses or medical conditions which would not permit the participant to be managed according to the protocol.
* Known hypersensitivity to the study drug(s) or their components.
* Prior CD19-directed CAR-T at any time, autologous hematopoietic cell transplantation within 6 weeks, or allogeneic hematopoietic cell transplantation within 3 months. Allogeneic hematopoietic cell transplantation recipients must be free of clinically-significant graft-versus-host disease (GvHD) and must be off immunosuppression for GvHD for at least 4 weeks before enrollment.
* Untreated and/or uncontrolled cardiovascular conditions and/or symptomatic cardiac dysfunction (including cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects) or unstable angina congestive heart failure or myocardial infarction within the previous year.
* Active, uncontrolled bacterial, fungal, or viral infection within 14 days prior to enrollment
* Pregnant or breastfeeding women.
* Inability to discontinue use of moderate or strong CYP3A inducers or inhibitors during the ramp-up treatment period with sonrotoclax.
* Live vaccination within 4 weeks prior to enrollment or who plan to receive a live vaccine during treatment or within 90 days post last dose.
* Inability to swallow capsules or tablets or have any diseases significantly affecting GI function
* Active central nervous system (CNS) disease; Participants with stable CNS disease are eligible.
* Growth factors within 28 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response post CAR-T | 3.5 years

SECONDARY OUTCOMES:
Objective Response Rate assessed by the Lugano Classification | 3.5 years
1 year Progression-Free Survival | 4 years
Overall Survival | 4 years
Number and Severity of Adverse Events | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Diego Villa, Study Chair — BCCA-Vancouver Cancer Centre; Robert Puckrin, Study Chair — Tom Baker Cancer Centre, Calgary, AB Canada

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: As per CCTG policies
URL: https://www.ctg.queensu.ca/public/policies